CLINICAL TRIAL: NCT00722267
Title: Patient Perception of Symptom Variability. A Cross-sectional Study of Patients With Severe COPD.
Brief Title: European Non-interventional Study in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Rick Lones, MD, European Medical Affairs Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-REU-DUM-2007/1
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2009-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: severe COPD; COPD symptoms; variability of symptoms; patient's perception
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is investigating how patients with severe stable state COPD perceive the variability of their symptoms throughout the day, the week and the year; the impact of these variations on their daily activities or sleep quality and how they deal with their treatments. For this purpose patients will be asked to answer a questionnaire over the phone

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of COPD
* FEV1<50% and FEV1/FVC<0.7 according to lung function data in medical records.
* Smoker or ex-smoker > 10 pack-years
* Informed consent obtained

Exclusion Criteria:

* Ongoing exacerbation of COPD or within the previous 3 months
* Any other significant respiratory disease (including asthma and allergic rhinitis)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating physicians (GPs and Respiratory physicians) will be asked to recruit 4 patients (on average). The first patients presenting for a consultation for any reason, who meet eligibility criteria, and give informed consent, should be enrolled.
Sampling Method: Probability Sample
Enrollment: 7400 (Estimated)
Dates: Start 2008-07; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Patient's perception of the variability of symptoms due to severe stable state COPD throughout the day, the week and the year | Once

SECONDARY OUTCOMES:
Impact of symptoms (and variability of symptoms) on the patient's morning & daily living activities and sleep quality. | Once
Describe how patient use their COPD treatment | Once
Factors that may influence the patient's perception of symptom variability | Once

CONTACTS AND LOCATIONS:
Locations (606):
- Austria (18):
  - Research Site, Baden
  - Research Site, Feldbach
  - Research Site, Feldkirch
  - Research Site, Güssing
  - Research Site, Innsbruck
  - Research Site, Landeck
  - Research Site, Linz
  - Research Site, Linz-Urfahr
  - Research Site, Neusiedl am See
  - Research Site, Salzburg
  - Research Site, Schlüsslberg
  - Research Site, Steyr
  - Research Site, Thalheim/Wels
  - Research Site, Vienna
  - Research Site, Wels
  - Research Site, Winden
  - Research Site, Wr.Neustadt
  - Research Site, Zwettl Stadt
- Belgium (34):
  - Research Site, Aalst
  - Research Site, Antwerp
  - Research Site, Ath
  - Research Site, Bertogne
  - Research Site, Boussu
  - Research Site, Carnières
  - Research Site, Châtelet
  - Research Site, Courcelles
  - Research Site, Duffel
  - Research Site, Florennes
  - Research Site, Geraardsbergen
  - Research Site, Ghent
  - Research Site, Gosselies
  - Research Site, Haine-Saint-Paul
  - Research Site, Houthulst
  - Research Site, Houtvenne
  - Research Site, Izegem
  - Research Site, Kortessem
  - Research Site, Kraainem
  - Research Site, Lauwe
  - Research Site, Liège
  - Research Site, Lokeren
  - Research Site, Lommel
  - Research Site, Micheroux
  - Research Site, Mons
  - Research Site, Montzen
  - Research Site, Olsene
  - Research Site, Ostend
  - Research Site, Saive
  - Research Site, Schaarbeek
  - Research Site, Vielsalm
  - Research Site, Willebroek
  - Research Site, Woluwe-Saint-Pierre - Sint-Pieters-Woluwe
  - Research Site, Zomergem
- Denmark (21):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Brørup
  - Research Site, Copenhagen S
  - Research Site, Elsinore
  - Research Site, Frederikssund
  - Research Site, Fredriksberg
  - Research Site, Grenå
  - Research Site, Holbæk
  - Research Site, Holstebro
  - Research Site, Hvidovre
  - Research Site, Ikast
  - Research Site, Jægerspris
  - Research Site, Middelfart
  - Research Site, Oksbøl
  - Research Site, Præstø
  - Research Site, Roskilde
  - Research Site, Sindal
  - Research Site, Skive
  - Research Site, Svinninge
  - Research Site, Thisted
- Finland (20):
  - Research Site, Ekenäs
  - Research Site, Hämeenlinna
  - Research Site, Helsingin Kaupunki
  - Research Site, Jakobstad
  - Research Site, Kajaani
  - Research Site, Klaukkala
  - Research Site, Kuopio
  - Research Site, Lahti
  - Research Site, Lappeenranta
  - Research Site, Lohja
  - Research Site, Mikkeli
  - Research Site, Närpes
  - Research Site, Oulu
  - Research Site, Pori
  - Research Site, Pyhäjoki
  - Research Site, Sairaalamaki
  - Research Site, Seinäjoki
  - Research Site, Tampere
  - Research Site, Turku
  - Research Site, Vääksy
- France (161):
  - Research Site, Agde
  - Research Site, Aix-en-Provence
  - Research Site, Albi
  - Research Site, Amélie-les-Bains
  - Research Site, Angers
  - Research Site, Annecy
  - Research Site, Argentan
  - Research Site, Arles
  - Research Site, Armentiere
  - Research Site, Auchy-les-Mines
  - Research Site, Augny
  - Research Site, Aureilhan
  - Research Site, Avignon
  - Research Site, Babarthe Sur Leze
  - Research Site, Bandol
  - Research Site, Bar-le-Duc
  - Research Site, Bayonne
  - Research Site, Beauvais
  - Research Site, Belfort
  - Research Site, Béthune
  - Research Site, Béziers
  - Research Site, Bois-Guillaume
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Castelnau-le-Lez
  - Research Site, Castelnaudary
  - Research Site, Cerizay
  - Research Site, Chalon En Champagne
  - Research Site, Champs-sur-Marne
  - Research Site, Charleville-Mézières
  - Research Site, Châteauroux
  - Research Site, Clermont-Ferrand
  - Research Site, Colmar
  - Research Site, Colomiers
  - Research Site, Corbeil Essones
  - Research Site, Creil
  - Research Site, Créteil
  - Research Site, Croix
  - Research Site, Cugnaux
  - Research Site, Cuise-la-Motte
  - Research Site, Denain
  - Research Site, Desseges
  - Research Site, Draguignan
  - Research Site, Échirolles
  - Research Site, Épernay
  - Research Site, Épinal
  - Research Site, Férolles-Attilly
  - Research Site, Foix
  - Research Site, Fontainebleau
  - Research Site, Forbach
  - Research Site, Giens
  - Research Site, Gonesse
  - Research Site, Grasse
  - Research Site, Graulhet
  - Research Site, Guingamp
  - Research Site, Harnes
  - Research Site, Hyères
  - Research Site, Istres
  - Research Site, Juan-les-Pins
  - Research Site, La Baule-Escoublac
  - Research Site, La Destrousse
  - Research Site, La Grande-Motte
  - Research Site, La Rochelle
  - Research Site, Laon
  - Research Site, Laval
  - Research Site, Le Brusc
  - Research Site, Le Chesnay
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Perreux-sur-Marne
  - Research Site, Liévin
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lomme
  - Research Site, Lourdes
  - Research Site, Lucé
  - Research Site, Lyon
  - Research Site, Mamande
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Marseille
  - Research Site, Maury
  - Research Site, Maxéville
  - Research Site, Mensignac
  - Research Site, Molsheim
  - Research Site, Mont-de-Marsan
  - Research Site, Montauban
  - Research Site, Montbéliard
  - Research Site, Montfermeil
  - Research Site, Montigny-lès-Metz
  - Research Site, Morlaix
  - Research Site, Nantes
  - Research Site, Nevers
  - Research Site, Nice
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Nogent-sur-Marne
  - Research Site, Obernai
  - Research Site, Olioules
  - Research Site, Orsay
  - Research Site, Paris
  - Research Site, Perpignan
  - Research Site, Pertuis
  - Research Site, Pierre-Bénite
  - Research Site, Plouzané
  - Research Site, Poitiers
  - Research Site, Pont-Évêque
  - Research Site, Pontallier Sur Saone
  - Research Site, Ponteil Et Bresis
  - Research Site, Quimper
  - Research Site, Quincy-Voisins
  - Research Site, Remiremont
  - Research Site, Renazé
  - Research Site, Rennes
  - Research Site, Roanne
  - Research Site, Rochefort
  - Research Site, Ronchin
  - Research Site, Rougegoutte
  - Research Site, Royan
  - Research Site, Rueil-Malmaison
  - Research Site, Saint Aubin Des Chateux
  - Research Site, Saint Feyre
  - Research Site, Saint-Amand-les-Eaux
  - Research Site, Saint-Aubin-lès-Elbeuf
  - Research Site, Saint-Cyr-sur-Loire
  - Research Site, Saint-Dié
  - Research Site, Saint-Etienne
  - Research Site, Saint-Genis-Laval
  - Research Site, Saint-Hilaire Agen
  - Research Site, Saint-Jean-d'Angély
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Julien-en-Genevois
  - Research Site, Saint-Mamert-du-Gard
  - Research Site, Saint-Mandrier-sur-Mer
  - Research Site, Saint-Michel-sur-Orge
  - Research Site, Saint-Priest
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Saint-Quentin
  - Research Site, Saint-Romain-la-Motte
  - Research Site, Saint-Rome-de-Cernon
  - Research Site, Saint-Symphorien-sur-Coise
  - Research Site, Saintes
  - Research Site, Salomé
  - Research Site, Saulnes
  - Research Site, Segré
  - Research Site, Sélestat
  - Research Site, Soissons
  - Research Site, Ste Severe Sur Indre
  - Research Site, Strasbourg
  - Research Site, Taden
  - Research Site, Tarbes
  - Research Site, Thionville
  - Research Site, Toul
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Vabres Labaye
  - Research Site, Vannes
  - Research Site, Venerque
  - Research Site, Verdun
  - Research Site, Vénissieux
  - Research Site, Villefranche
- Germany (88):
  - Research Site, Arnsberg
  - Research Site, Augsburg
  - Research Site, Bad Krozingen
  - Research Site, Bad Sooden-Allendorf
  - Research Site, Bad Vilbel
  - Research Site, Belm
  - Research Site, Bergisch Gladbach
  - Research Site, Berlin
  - Research Site, Bernau
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Borchen
  - Research Site, Borstel
  - Research Site, Brakel
  - Research Site, Burkhardtsdorf
  - Research Site, Castrop-Rauxel
  - Research Site, Cologne
  - Research Site, Delitzsch
  - Research Site, Dieburg
  - Research Site, Dreieich
  - Research Site, Dresden
  - Research Site, Eckental
  - Research Site, Elbingerode
  - Research Site, Eschwege
  - Research Site, Essen
  - Research Site, Frankenberg
  - Research Site, Frankfurt
  - Research Site, Franzburg
  - Research Site, Freiburg im Breisgau
  - Research Site, Freital
  - Research Site, Friedrichsthal
  - Research Site, Fürstenfeldbruck
  - Research Site, Fürth
  - Research Site, Gelnhausen
  - Research Site, Gelsenkirchen
  - Research Site, Gerolzhofen
  - Research Site, Haan
  - Research Site, Halle
  - Research Site, Haltern
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Hemmingen
  - Research Site, Ingolstadt
  - Research Site, Kamen
  - Research Site, Kempten
  - Research Site, Kiel
  - Research Site, Köthen
  - Research Site, Kronach
  - Research Site, Laichingen
  - Research Site, Leinach
  - Research Site, Leipzig
  - Research Site, Leopoldshöhe
  - Research Site, Liebenau
  - Research Site, Lüdenscheid
  - Research Site, Magdeburg
  - Research Site, Mammendorf
  - Research Site, Manching
  - Research Site, Marburg
  - Research Site, Marktheidenfeld
  - Research Site, Moers
  - Research Site, Mühlhausen
  - Research Site, Niesky
  - Research Site, Nuremberg
  - Research Site, Oranienburg
  - Research Site, Osnabrück
  - Research Site, Pfronten
  - Research Site, Pleystein
  - Research Site, Pocking
  - Research Site, Potsdam
  - Research Site, Puchheim
  - Research Site, Roth
  - Research Site, Ruhmannsfelden
  - Research Site, Saarbrücken
  - Research Site, Saerbeck
  - Research Site, Schwabach
  - Research Site, Schwedt
  - Research Site, Sebnitz
  - Research Site, Solingen
  - Research Site, Starzach
  - Research Site, Straubing
  - Research Site, Stuttgart
  - Research Site, Teterow
  - Research Site, Welver
  - Research Site, Westerland
  - Research Site, Wettin
  - Research Site, Wiesbaden
  - Research Site, Witten
  - Research Site, Zerbst
- Greece (20):
  - Research Site, Athens
  - Research Site, Chalcis
  - Research Site, Chania
  - Research Site, Drapetsona
  - Research Site, Florina
  - Research Site, Heraklio
  - Research Site, Ilioúpoli
  - Research Site, Itháki
  - Research Site, Kalamaria
  - Research Site, Kifissia
  - Research Site, Koropí
  - Research Site, Lamia
  - Research Site, Messíni
  - Research Site, N.Santa
  - Research Site, Pátrai
  - Research Site, Platamonas
  - Research Site, Preveza
  - Research Site, Serres
  - Research Site, Thessaloniki
  - Research Site, Véroia
- Ireland (8):
  - Research Site, Cavan
  - Research Site, Dublin
  - Research Site, Enniscorthy
  - Research Site, Gorey
  - Research Site, Letterkenny
  - Research Site, Mullingar
  - Research Site, Turloughmore
  - Research Site, Waterford
- Italy (31):
  - Research Site, Alife
  - Research Site, Avezzano
  - Research Site, Badolato
  - Research Site, Balsorano
  - Research Site, Carsoli
  - Research Site, Casagiove
  - Research Site, Caserta
  - Research Site, Ceparana-Carpena
  - Research Site, Copertino
  - Research Site, Cutrofiano
  - Research Site, Eboli
  - Research Site, Grosseto
  - Research Site, La Spezia
  - Research Site, Macerata Campania
  - Research Site, Montiano
  - Research Site, Napoli
  - Research Site, Orbetello
  - Research Site, Ortonovo
  - Research Site, Paganico
  - Research Site, Palermo
  - Research Site, Pellezzano
  - Research Site, Pontecagnano
  - Research Site, Rispescia
  - Research Site, S.Maria Di Cantanzzaro
  - Research Site, Salerno
  - Research Site, San Felice A Cancello
  - Research Site, San Nicola la Strada
  - Research Site, San Pietro in Lama
  - Research Site, Srubo
  - Research Site, Trasacco
  - Research Site, Veglie
- Netherlands (29):
  - Research Site, 's-Hertogenbosch
  - Research Site, Almere Stad
  - Research Site, Alphen aan den Rijn
  - Research Site, Amsterdam
  - Research Site, Andijk
  - Research Site, Arnhem
  - Research Site, Delfzijl
  - Research Site, Den Helder
  - Research Site, Drachten
  - Research Site, Enschede
  - Research Site, Gouda
  - Research Site, Groningen
  - Research Site, Heemstede
  - Research Site, Heerlen
  - Research Site, Hilversum
  - Research Site, Hoogwoud
  - Research Site, Landgraaf
  - Research Site, Leiden
  - Research Site, Meppel
  - Research Site, Onstwedde
  - Research Site, Oude Pekela
  - Research Site, Roermond
  - Research Site, Rotterdam
  - Research Site, Sint Philipsland
  - Research Site, Sneek
  - Research Site, The Hague
  - Research Site, Tilburg
  - Research Site, Utrecht
  - Research Site, Zutphen
- Norway (6):
  - Research Site, Ålesund
  - Research Site, Brevik
  - Research Site, Hakadal
  - Research Site, Molde
  - Research Site, Oslo
  - Research Site, Trondheim
- Portugal (6):
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Melgaço
  - Research Site, Odivelas
  - Research Site, Santarém
  - Research Site, Torres Vedras
- Spain (82):
  - Research Site, A Coruña
  - Research Site, Alamagro
  - Research Site, Alcal de Henares
  - Research Site, Alcoy
  - Research Site, Alicante
  - Research Site, Andújar
  - Research Site, Arcos de La Fortera
  - Research Site, As Pontes de García Rodríguez
  - Research Site, Avilés
  - Research Site, Ávila
  - Research Site, Badalona
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Bellaterra
  - Research Site, Bilbao
  - Research Site, Boqueixon (Pontella)
  - Research Site, Brean Alta
  - Research Site, Burela de Cabo
  - Research Site, Burgos
  - Research Site, Burguillos
  - Research Site, Carvaca de La Cruz
  - Research Site, Castellon
  - Research Site, Cervera
  - Research Site, Cesuras
  - Research Site, Cuenca
  - Research Site, Donostia / San Sebastian
  - Research Site, El Vendrell
  - Research Site, Ferrol
  - Research Site, Fuenlabrada
  - Research Site, Girona
  - Research Site, Granollers
  - Research Site, Guadalajara
  - Research Site, Huelva
  - Research Site, Jaén
  - Research Site, Joiosa
  - Research Site, La Almunia de Doña Godina
  - Research Site, Laredo
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Leganés
  - Research Site, Llobregat
  - Research Site, Logroño
  - Research Site, Lora del Río
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Manacor
  - Research Site, Melilla
  - Research Site, Mieres
  - Research Site, Montilla
  - Research Site, Murcia
  - Research Site, Outes
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Ponferrada
  - Research Site, Porreres
  - Research Site, Portugalete
  - Research Site, Pozoblanco
  - Research Site, Quart de Poblet
  - Research Site, Quintanar del Rey
  - Research Site, Ronda
  - Research Site, Sabadell
  - Research Site, Sagunto
  - Research Site, Salamanca
  - Research Site, Salt
  - Research Site, San Vicent del Raspeig
  - Research Site, Sant Antoni de Portmany
  - Research Site, Sant Boi de Llobregat
  - Research Site, Sant Pere de Ribes
  - Research Site, Santa Coloma de Gramenet
  - Research Site, Santa Coloma de Queralt
  - Research Site, Santiago de Compostela
  - Research Site, Santurtzi
  - Research Site, Teruel
  - Research Site, Toledo
  - Research Site, Torrebonica
  - Research Site, Torrelavega
  - Research Site, Valdepeñas
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Vigo
  - Research Site, Viladecans
  - Research Site, Xàtiva
- Sweden (22):
  - Research Site, Angered
  - Research Site, Åtvidaberg
  - Research Site, Bjärred
  - Research Site, Borlänge
  - Research Site, Danderyd
  - Research Site, Falun
  - Research Site, Forserum
  - Research Site, Fredriksberg
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Höllviken
  - Research Site, Hunnebostrand
  - Research Site, Kälarne
  - Research Site, Kinna
  - Research Site, Kungsbacka
  - Research Site, Malmo
  - Research Site, Norrköping
  - Research Site, Östersund
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Uppsala
  - Research Site, Värnamo
- Switzerland (8):
  - Research Site, Bern
  - Research Site, Herisau
  - Research Site, Lausanne
  - Research Site, Martigny-Ville
  - Research Site, Samedan
  - Research Site, Spiez
  - Research Site, Wolfgang
  - Research Site, Zurich
- Turkey (Türkiye) (22):
  - Research Site, Adana
  - Research Site, Akyokus-Konya
  - Research Site, Anamur/mersin
  - Research Site, Ankara
  - Research Site, Aydin
  - Research Site, Denizli
  - Research Site, Erzincan
  - Research Site, Eskişehir
  - Research Site, Hatay
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, K.Maras
  - Research Site, Konya
  - Research Site, Malatya
  - Research Site, Mezitli-Mersin
  - Research Site, Osmaniye
  - Research Site, Sakarya
  - Research Site, Sanliurfa
  - Research Site, umraniye-Istanbul
  - Research Site, Yenişehir
  - Research Site, Yozgat
  - Research Site, Zonguldak
- United Kingdom (30):
  - Research Site, Ashwell
  - Research Site, Atherstone
  - Research Site, Barry
  - Research Site, Birmingham
  - Research Site, Blackburn
  - Research Site, Blackpool
  - Research Site, Bradford-on-Avon
  - Research Site, Cardiff
  - Research Site, Chertsey
  - Research Site, Chesterfield
  - Research Site, Chippenham
  - Research Site, Cookstown
  - Research Site, Corsham
  - Research Site, Coventry
  - Research Site, Doncaster
  - Research Site, Fife
  - Research Site, High Valleyfield
  - Research Site, Maidenhead
  - Research Site, Nottingham
  - Research Site, Peterborough
  - Research Site, Plymouth
  - Research Site, Ruislip
  - Research Site, Sandy
  - Research Site, Southampton
  - Research Site, Sunbury-on-Thames
  - Research Site, Thornton Heath
  - Research Site, Trowbridge
  - Research Site, Warminster
  - Research Site, Wells-next-the-Sea
  - Research Site, Westbury

REFERENCES:
- [Derived] Kessler R, Partridge MR, Miravitlles M, Cazzola M, Vogelmeier C, Leynaud D, Ostinelli J. Symptom variability in patients with severe COPD: a pan-European cross-sectional study. Eur Respir J. 2011 Feb;37(2):264-72. doi: 10.1183/09031936.00051110. Epub 2010 Nov 29. PMID 21115606